CLINICAL TRIAL: NCT03665519
Title: Clinical Trial on the Effect of Sublimated Mare Milk Supplement in Patients With Biliary Cholangitis
Brief Title: Clinical Trial on the Effect of the Sublimated Mare Milk Supplement on Primary Biliary Cholangitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Scientific Medical Center, Kazakhstan (Other Government)
Collaborators: Eurasia Invest Ltd. (Industry); Ministry of Education and Science, Republic of Kazakhstan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NNMC.MM.BC.01
Record Dates: First submitted 2018-09-06; First posted 2018-09-11 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Primary Biliary Cirrhosis; Primary Biliary Cholangitis; Mare Milk
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement and ursodeoxycholic acid therapy. (Experimental): Participants will take a supplement (sublimated mare milk) of 1 sachet (20 mg) dissolved in 200 ml of warm water (36-37 °C) twice/day accompanied with standard therapy of ursodeoxycholic acid therapy (dosage of 15/kg/day) for 3 months.
  Interventions: Dietary Supplement: Sublimated mare milk; Drug: Ursodeoxycholic Acid
- Ursodeoxycholic acid therapy only. (Other): Patients would be given the standard treatment of ursodeoxycholic acid only for 3 months.
  Interventions: Drug: Ursodeoxycholic Acid

INTERVENTIONS:
Dietary Supplement: Sublimated mare milk — The dietary supplement mare milk product, which is obtained from fresh mare milk (few hours) through sublimation process.
  Arms: Dietary supplement and ursodeoxycholic acid therapy.
Drug: Ursodeoxycholic Acid — Ursodeoxycholic acid treatment will be given for 3 months.

SUMMARY:
This study evaluates the effect of sublimated mare milk supplement on patients with biliary cholangitis

DETAILED DESCRIPTION:
Primary biliary cholangitis, formerly known as primary biliary cirrhosis, is a rare chronic disease that primarily affects women. Primary biliary cholangitis often progresses to the terminal stage of liver cirrhosis with its inherent complications. At this stage, the only way to save the patient's life is liver transplantation, and is accompanied by a number of painful symptoms (itching, mucous dryness, abdominal discomfort, fatigue), often restless legs syndrome, insomnia, depression and cognitive dysfunction.

The goal of the treatment is to prevent the terminal stage of cirrhosis of the liver and to alleviate the accompanying symptoms. Conventional drug therapy is aimed at slowing the progression of the disease and includes both approved for the use of these medications (ursodeoxycholic acid) and used outside the approved indications (derivatives of fibric acid, budesonide).

The role of this clinical trial is to increase the effectiveness of therapy for this disease. Against the background of the complexity of the treatment of primary biliary cholangitis, clinical medicine acquires a remedy in the form of a natural product - mare's milk, preventive, dietary, medicinal effects of which have been known for a long time. There are data from studies that have shown the efficacy and safety of using mare milk in patients with atopic dermatitis as well as with inflammatory bowel diseases. For the liver diseases, there are no reported studies.

In this trial, there will be two parallel groups: Interventional (supplement with standard treatment first for 3 months) and Standard treatment group. Differences in clinical, laboratory, liver encephalopathy and asthenia will be evaluated between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with morphologically verified diagnosis of primary biliary cholangitis
* Aged 18 to 75 years
* Willingness to consent to participate in the study
* Consent to adhere to treatment

Exclusion Criteria:

* Alcohol and/or drug dependence
* Presence of liver cirrhosis class C based on Child Pugh classification
* Allergic reaction to dairy products
* Presence of mental diseases, severe concomitant pathology
* Pregnancy and/or lactation
* Lactose intolerance
* Refusal to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Biochemical changes in liver function. | Baseline, Month 4
  Levels of alanine aminotransferase and aspartate aminotransferase will be measured from a biochemical blood test.
Change in intensity of asthenia in patients. | Baseline, Month 4
  Intensity of asthenia will be assessed with the State-Asthenic Scale by L. Malkova (adapted by Chertova) with scores less than 50 and more than 100 indicating no asthenia and pronounced asthenia respectively.
Evaluation of liver histology. | Month 4
  Liver histology, histochemistry, immunohistochemistry will be evaluated based on biopsy samples.
Change from baseline in hepatic encephalopathy indicator. | Baseline, Month 4
  Presence and stage of hepatic encephalopathy will be determined using the Reitan test (number connection test)

SECONDARY OUTCOMES:
Change in inflammatory biomaker (erythrocyte sedimentation rate). | Baseline, Month 4
  The erythrocyte sedimentation rate will be measured using the Panchenkov method
Determination of cholestasis presence/stage. | Baseline, Month 4
  Cholestasis will be assessed according to levels of gamma-glutamyltransferase, Alkaline phosphatase, direct bilirubin, total bilirubin from blood samples.
Evaluation of changes in synthetic function of liver (prothrombin time). | Baseline, Month 4
  Synthetic function of liver will be evaluated from the blood test result of prothrombin time.
Evaluation of changes in synthetic function of liver (fibrinogen). | Baseline, Month 4
  Synthetic function of liver will be evaluated from blood test results of fibrinogen, and platelet count.
Evaluation of changes in synthetic function of liver (albumin). | Baseline, Month 4
  Synthetic function of liver will be evaluated from blood test results of albumin.
Evaluation of changes in low-density lipoprotein. | Baseline, Month 4
  Synthetic function of liver will be evaluated from blood test results of low-density lipoprotein.
Evaluation of changes in total protein. | Baseline, Month 4
  Synthetic function of liver will be evaluated from blood test results of total protein.
Evaluation of changes in platelet count. | Baseline, Month 4
  Synthetic function of liver will be evaluated blood test results of platelet count.
Detection of anemia. | Baseline, Month 4
  Blood hemoglobin level will be used as a parameter for diagnosing anemia.
Hepatic hypertension | Baseline, Month 4
  Detection of hepatic hypertension will be carried out via platelet level assessment from the blood samples.

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Medical Center, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foekel C, Schubert R, Kaatz M, Schmidt I, Bauer A, Hipler UC, Vogelsang H, Rabe K, Jahreis G. Dietetic effects of oral intervention with mare's milk on the Severity Scoring of Atopic Dermatitis, on faecal microbiota and on immunological parameters in patients with atopic dermatitis. Int J Food Sci Nutr. 2009;60 Suppl 7:41-52. doi: 10.1080/09637480802249082. Epub 2009 May 21. PMID 19462320
- [Background] Guri A, Paligot M, Crevecoeur S, Piedboeuf B, Claes J, Daube G, Corredig M, Griffiths MW, Delcenserie V. In vitro screening of mare's milk antimicrobial effect and antiproliverative activity. FEMS Microbiol Lett. 2016 Jan;363(2):fnv234. doi: 10.1093/femsle/fnv234. Epub 2015 Dec 9. PMID 26656278
- [Background] Valiev AG, Valieva TA, Valeeva GR, Speranskii VV, Levachev MM. [The effect of the essential fatty acids in mare's milk on the function of the immune system and of nonspecific resistance in rats]. Vopr Pitan. 1999;68(3):3-6. Russian. PMID 10392421
- [Background] Wulijideligen, Asahina T, Hara K, Arakawa K, Nakano H, Miyamoto T. Production of bacteriocin by Leuconostoc mesenteroides 406 isolated from Mongolian fermented mare's milk, airag. Anim Sci J. 2012 Oct;83(10):704-11. doi: 10.1111/j.1740-0929.2012.01010.x. Epub 2012 Mar 13. PMID 23035710
- See also: Dietetic Efficacy of Mare's Milk for Patients With Chronic Inflammatory Bowel Diseases — https://clinicaltrials.gov/ct2/show/NCT00940576